CLINICAL TRIAL: NCT06116071
Title: Pilot Study to Assess Immune Biomarkers and Growth Factors Related to Bone Pathology in Pediatric Patients With Gaucher Disease
Brief Title: Biomarkers Related to Bone in Pediatric Gaucher Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 23-LDRTC-02
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-10

CONDITIONS: Gaucher Disease; Bone Diseases
MeSH Terms: conditions — Gaucher Disease; Bone Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GD subjects with normal growth rate and no bone involvement: No drug interventions.
- GD type 1 subjects with evidence of bone involvement: No drug interventions.
- GD type 3 subjects: No drug interventions.
- Non-GD age and gender-matched controls with normal growth rate and no known bone complications: No drug interventions.

SUMMARY:
Aims of the observational study is to establish novel blood-based biomarkers for grading bone disease in pediatric patients with Gaucher disease (GD). Patients with clinically confirmed GD: deficient GCase enzyme activity and corresponding genetic analysis will be eligible for enrollment. Levels of Lyso-Gb1, chitotriosidase, and CCL18 will be established for future bone biomarkers correlation analysis. Skeletal involvement will be assessed using standard clinical diagnostic tools, such as skeletal radiology and/or (DEXA). The comparator group will include age-matched healthy controls.

Clinically confirmed patients with GD will be stratified based on their disease severity (Gaucher disease type 1 and Gaucher disease type 3) and bone pathology findings. In addition, given that growth is a dynamic process during the pediatric age group, results will be ascertained with respect to phases of growth, i.e., early childhood, late childhood, adolescent, and young adult age groups. At the conclusion of the study, investigatirs expect to establish specific biomarkers of bone development and pathology in pediatric GD patients.

DETAILED DESCRIPTION:
Gaucher disease (GD), the most common lysosomal storage disorder, is caused by a deficiency of the enzyme glucocerebrosidase. Clinically, there are three sub-types according to neurological involvement. Type 1 GD (GD1) is non-neuronopathic GD, and GD types 2 and 3 (GD2-3) are neuronopathic forms. Bone involvement includes skeletal structural abnormalities such as Erlenmeyer flask deformities, cystic changes, growth retardation, progressive kyphoscoliosis, osteonecrosis, bone density abnormalities, bone fragility, and pathological fractures occur at a spectrum in different GD clinical types.

While bone crises are rare (often referred to as Gaucher crises), avascular necrosis (AVN) may occur in the pediatric age group with long-term morbidity and is often associated with chronic pain and orthopedic deformities requiring multiple surgical interventions.

As known, the development of the skeleton development (longitudinal and bone mass growth) is subject to both environmental and genetic influences. During childhood, skeletal growth is characterized by rapid bone growth and continues to lengthen bones by adding bone tissue on the epiphyseal plate until adolescence. The thickening of long bones is processed by adding bony tissue to its surface. The process of bone remodeling and repair continues after birth and adulthood.

Bone marrow infiltration and bone remodeling defects termed "Erlenmeyer flask deformity" are the most common GD-related bone diseases. Without intervention directed at GD, bone involvement usually starts before puberty. Moreover, children with severe GD present retarded growth and delayed puberty (<5th percentile in 34% of children). However, the underlying mechanisms of regulation of bone development and related complications in the pediatric age group in GD are not yet fully known. Neither the bone-specific biomarkers nor their relationship regarding growth factors associated with normal bone turnover during the normal growth process have been studied in detail in GD in the pediatric age group. Abnormalities in skeletal growth and bone turnover may be related to the abnormal regulation of some growth factors, for example, the elevation of fibroblast growth factor 23 (FGF23) or inhibition of insulin-like growth factors (IGFs) resulting in bone growth impartment. Moreover, chronic inflammation leads to alterations in the function and differentiation of osteoclasts and osteoblasts, which participate in bone growth and remodeling.

Furthermore, the evaluation of bone involvement could be challenging for the pediatric age group. The marrow replacement due to GD that moves in the opposite direction with the expected disappearance of the red marrow makes it challenging to evaluate the bone marrow using MRI and requires experience and technical skills to interpret the imaging studies. In addition, the technique of bone density evaluation is still not uniform in children, especially for different age groups.

ELIGIBILITY:
Inclusion Criteria:

1. The parent or legal guardian and the participant who is eligible to provide assent are able and willing to provide informed consent and assent when applicable.
2. The participant is 5-21 years of age at the initial visit.
3. The participant has a confirmed diagnosis of GD type 1 or type 3 (biochemically and/or genetically).
4. In the investigator's opinion, the subject is capable of understanding and complying with protocol requirements.
5. The subject or, when applicable, the subject's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. Any subject who does not meet any of the following criteria will not qualify for the study.
2. Any current active chronic infection such as HIV, Hepatitis B or C.
3. Pregnancy or breastfeeding for females.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with clinically confirmed GD: deficient GCase enzyme activity and corresponding genetic analysis will be eligible for enrollment. GD patients with and without bone abnormalities and growth retardation. The study population will comprise patients with Gaucher disease from Lysosomal & Rare Disorders Research & Treatment Center and who were referred to Lysosomal & Rare Disorders Research & Treatment Center who are 21 years or younger.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood-based biomarkers that correlate with bone involvement in pediatric patients with GD. | 24 months
  DMP-1, Osteocalcin, DKK-1, BAP, RANKL, OPG, TRAP5b, CTX, SOST, SFRP1, PICP,PINP, CCL1, GM-CSF, Il-4, Il-5, Il-6, Il-10, TNFalpha concentrations units/ml
Plasma Growth factors and bone development, including bone age, skeletal maturation and bone development abnormalities | 24 months
  IGF-1, IGFBP-3, TGFbeta, BMP6, BMP9, FGF2, FGF18, FGF21, FGF23 concentration in plasma units/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — Lysosomal and Rare Disorders Research and Treatment Center
Locations (1):
- Lysosomal and Rare disorder research and treatment center, Fairfax, Virginia, United States